CLINICAL TRIAL: NCT00277615
Title: Clinical Evaluation of a Portable Ultrasound Bladder Scanner for Continuous Monitoring of Bladder Function in Children.
Brief Title: Evaluation Study of Ultrasound Bladder Scanner for Monitoring Bladder Function
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: SHUL2006; 2005-41-5570, 20050083
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Dysfunction of the Urinary Bladder
Keywords: Children; Bladder volume; Ultrasound

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate a novel ultrasound bladder scanning device designed particularly for children in children with bladder dysfunction.

DETAILED DESCRIPTION:
A continuous precise monitoring of bladder volume is of great impotence in many nephro-urological diseases in children.

Some children suffer from bladder dysfunctions that necessitate bladder emptying by catheterization. The bladder catheterizations are at present performed at fixed time intervals and are not based on the amount of urine in the bladder.

In order to avoid overfilling of the bladder, the interval between the emptying is set with a safety margin. This leads to at least some needless catheterizations and hereby discomfort for the children. A portable bladder monitor could possible give a measurement of the degreed of bladder filling and hereby minimize the number of catheterizations needed.

Another group of children suffers from daytime urinary incontinence as a result of overactive bladder syndrome. Home recordings of fluid intake and micturations are used for diagnosing the cause of the decease however; a portable bladder monitor system would possibly give a more true reflection of the bladder function.

With a prevalence of about 10 % nocturnal enuresis is the most common nephro-urological disorder of childhood. In this group of children a portable bladder monitor may enable a more precise measure of bladder function. In addition to this the monitor may be used as a alarm device in the treatment of the disorder.

The portable ultrasound bladder scanner tested has been designed particularly for children.

Hypothesis:

* The bladder volume estimated by the portable ultrasound bladder scanner is concordant with "true" bladder volume measured by catheterization in children.
* The portable ultrasound bladder scanner can be used for continuous non-invasive monitoring of bladder volume during natural fill in children with bladder dysfunction.

  30 children that suffer from bladder dysfunction and perform bladder emptying by catheterization will be recruited from the Center of Child Incontinence, Skejby University Hospital, Aarhus, Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4-16 yrs
* Dependent on bladder emptying by catheterization
* Informed consent

Exclusion Criteria:

* Wounds, scar tissue or staples in the suprapubic area
* Severe urinary incontinence

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with OAB
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2005-10; Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Hagstroem, MD, Principal Investigator — University of Aarhus
Locations (1):
- Department of pediatrics, University hospital of Aarhus, Skejby Sygehus, Aarhus, Aarhus N, Denmark